CLINICAL TRIAL: NCT00847496
Title: The Treatment of Partial Thickness Burns: Awbat(r) Versus Biobrane(r)
Brief Title: Awbat Versus Biobrane in Partial Thickness Burns
Acronym: Awbat
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Company went out of business
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-333; NCT00793533 (obsolete NCT alias)
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Burns
Keywords: Partial Thickness burn; Biological Dressing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AWBAT
  Interventions: Device: AWBAT
- 2 (Active Comparator): BIOBRANE(R)
  Interventions: Device: Biobrane

INTERVENTIONS:
Device: AWBAT — One-time application of dressing over partial-thickness burns
  Arms: 1
Device: Biobrane — One-time application over partial-thickness burns
  Arms: 2

SUMMARY:
• To determine if AWBAT, used in treating partial-thickness burns, would provide better healing, pain control, control of infection, shorter length of hospital stay, lower costs, and improved scarring and long term recovery when compared to Biobrane®.

DETAILED DESCRIPTION:
Currently there is no "best covering" or a standard "approved care" for treating partial thickness burns. Several options are available; however, they all have shortcomings. The application of topical antimicrobial dressings is time consuming and the regular dressing changes often associated with pain. Homograft or cadaver skin is often unavailable or in great shortage for skin transplants. Biobrane®, a biosynthetic wound dressing constructed of a silicone film with a nylon fabric partially imbedded into the film, has been available and used at our institute for many years as a skin substitute. It has been shown to reduce pain and the number of necessary dressing changes, and significantly reduced healing time (1). Its main side effects, although rare, are the occasional occurrence of infections and allergic reactions to the material.

Recently, a new product, AWBAT, has been developed for the coverage of partial thickness burns. AWBAT is similar to Biobrane® in terms of silicone membrane thickness, the structure of nylon fabric that gives the dermal substitute its strength, and the use of collagen peptides on the inner side of the membrane. These peptides are used for the purpose of reacting with the fibrin in the wound in order to achieve good initial adherence and to accelerate re-epithelialization. The key novelties of AWBAT are the different pore size and modality of collagen peptide attachments. These two key modifications aim at a reduction of the above mentioned adverse reactions.

The purpose of this study is to compare AWBAT to Biobrane® for covering partial thickness-burn injuries. We wish to determine if AWBAT, used in treating partial-thickness burns, would provide better healing, pain control, control of infection, shorter length of hospital stay, and improved scarring and long term recovery when compared to Biobrane®.

ELIGIBILITY:
Inclusion Criteria:

* Partial thickness burns between 4% and 40% Total Body Surface Area(TBSA)
* Full thickness burns not to exceed 10% TBSA,
* Age as specified

Exclusion Criteria:

* Full thickness burns that require immediate excision and grafting
* Known allergic reaction against Biobrane
* Chemical and electrical burns

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Time to complete Healing | 5 - 14 days post injury/membrane application

SECONDARY OUTCOMES:
Occurence of Infection | entire study period

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — Shriners Hospital for Children and University of Texas Medical Branch
Locations (1):
- Shriners Hospital for Children, Galveston, Texas, United States